CLINICAL TRIAL: NCT02157818
Title: A Comparison of Dexmedetomidine Versus Midazolam for Conscious Sedation During Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS-TBNA)
Brief Title: A Comparison of Sedative Drugs for Conscious Sedation During Ultrasound Guided Transbronchial Needle Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jinwoo Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: dex512
Record Dates: First submitted 2014-06-01; First posted 2014-06-06 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Endobronchial Ultrasound Guided Transbronchial Needle Aspiration
MeSH Terms: interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midazolam (Active Comparator): midazolam IV bolus 0.05ml/kg bolus in 1minute. rescue drug(Midazolam) 1 mg, IV boluses for double blinding setting, we use saline, 0.4 mcg/kg IV bolus in 10 minutes and 0.5 mcg/kg/h, as placebo.
  Interventions: Drug: midazolam
- Dexmedetomidine (Experimental): Dexmedetomidine 0.4 mcg/kg IV bolus in 10 minutes. Dexmedetomidine 0.25-0.75 mcg/kg/h for RSS 3-5. Midazolam 1mg bolus IV pro re nata (PRN).
  for double blinding setting, IV bolus 0.05ml/kg bolus in 1minute.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: midazolam
  Arms: midazolam
Drug: Dexmedetomidine
  Arms: Dexmedetomidine

SUMMARY:
1. Appropriate sedation is needed for medical diagnosis, treatment, and the safety for patients. In non-surgical approaches, benzodiazepines are broadly used for ideal sedated status for patients.

   * However, especially in bronchoscope procedure, continuous monitoring of oxygen saturation is needed to prevent hypoxia due to respiratory distress induced by benzodiazepine.
   * A alpha-2 agonist, dexmedetomidine, which has similar sedative effect, but has less adverse effect of respiratory distress compared to previous agents, was introduced.
2. It is necessary to compare the efficacy and safety of dexmedetomidine with that of midazolam in ultrasound guided transbronchial needle aspiration (EBUS-TBNA).

   * Double blind randomized trial
   * Primary outcome: The number and duration of desaturation, volume of sedative, any use of rescue midazolam, and Ramsay Sedation Scale (RSS) score (for efficacy), and hypertension, tachycardia, any need for mandible support or manual ventilation, and any need for intubation (for safety).

ELIGIBILITY:
Inclusion Criteria:

* Patients who visit Seoul National University Hospital between 2014.04 - 2015.04
* Patients who undergo EBUS-TBNA during the period
* Aged between 18-75
* Patients who meet the criteria of American Society of Anesthesiologists (ASA) physical status classification I-III

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification >3
* Have glomerular filtration rate (GFR) less than 15ml/min 1.73m2 or undergoing hemodialysis
* End stage liver disease.
* Impaired ventricular functions (EF <30%)
* Patients with baseline oxygen desaturation (resting SpO2 <90%)
* Asthma or chronic obstructive pulmonary disease or a forced expiratory volume in 1 s (FEV1)of < 1.0 liter
* Bradycardia [baseline heart rate (HR)< 60 beats/min]
* Hypotension [baseline systolic arterial pressure (SAP) < 100 mm Hg]
* Pregnant state
* Those intolerant or with an allergy to the study drug
* those unable or who refused to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The number of Desaturation events | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room, an expected average of 2 hours
  The number of desaturation (SpO2 <90% for more than 5 seconds) events

SECONDARY OUTCOMES:
RSS score | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room, an expected average of 2 hours
  RSS score: at the beginning of the procedure, minimum RSS score, every 5 minute
Total dose of intratracheal lidocaine instillation | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room, an expected average of 2 hours
  Cumulative dose of lidocaine administered at bronchus by the endoscopist for local anesthesia by topical instillation.
  Topical lidocaine instillation is performed in both the two arms for procedure as routine bronchoscopy.
Endoscopist satisfaction | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room
  Endoscopist global satisfaction score based on a VAS score
Patient satisfaction | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room, an expected average of 2 hours
  Global patient satisfaction associated with the procedure. Score based on a VAS score measured before the patients leave the bronchoscopy room.
Use of rescue midazolam | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room, an expected average of 2 hours
  Use of rescue midazolam, total dose
Duration of desaturation (sec) | Patient followed for the entire duration of EBUS-TBNA, an expected average of 2 hours
Hemodynamic adverse event | Patient followed for the entire duration of EBUS-TBNA and until discharge of bronchoscopy room, an expected average of 2 hours
  Hypotension ( < mean BP 60 mmHg) Bradycardia ( < 50 bpm)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Choi SM, Park YS, Lee CH, Lee SM, Yoo CG, Kim YW, Lee J. Dexmedetomidine versus midazolam for sedation during endobronchial ultrasound-guided transbronchial needle aspiration: A randomised controlled trial. Eur J Anaesthesiol. 2021 May 1;38(5):534-540. doi: 10.1097/EJA.0000000000001370. PMID 33122573